CLINICAL TRIAL: NCT05131048
Title: Effects of Home-based Hip Strengthening Exercises on Pain, Range of Motion and Functional Disability in Knee Osteoarthritis Patients: a Randomized Controlled Trial
Brief Title: Home Based Hip Strengthening for Knee OA Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Faizan Asghar, Principal investigator, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 890-V
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis; home-based exercise plan; functional disability; obesity
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional group (Active Comparator): Patients will be given thermal therapy with the hot pack for 20 minutes followed by Conventional physiotherapy will consist of a set of exercises. The exercise components willl be chosen based on previous studies (Deyle 2000) and will comprises of
  * stretches of lower limb muscles (gastrocnemius, soleus and hamstring)
  * isometric quadriceps work
  * straight leg raising
  * Joint mobilization includes anteroposterior (AP) glide of the tibia on the femur
  * the patella glides in all directions Subjects will participate in a 45-minute physical therapy session, on alternate days weekly for 6 weeks, in our centre under the close surveillance of a physical therapist. A total of 24 sessions will be given to this group.
  Interventions: Other: conventional group
- interventional group (Experimental): Patients in this group will perform home-based hip Strengthening exercises to strengthen hip abductor and adductor muscles. Six different home-based exercises will be taught. This group will have 3 sessions in 1st week in the hospital under the supervision of a trained physiotherapist just to teach them and ensure that patients are doing exercises correctly on their own. After that, patients will perform exercises 5 days at home and 1 session at the hospital per week. The therapist will be trained to deliver different exercises and adjust the intensity of exercise accordingly advise the participants to complete 10 repetitions of every exercise at home96.
  * Abduction in side-lying
  * Abduction in standing
  * Standing wall isometric hip abduction
  * Hip Adduction in side-lying
  * Hip abduction in a standing position
  * Towel press
  Interventions: Other: experimental group

INTERVENTIONS:
Other: conventional group — this group will perform conventional therapy
  Arms: Conventional group
Other: experimental group — this group will perform home based exercises
  Arms: interventional group

SUMMARY:
In knee osteoarthritis patients, weakness of hip abductor muscles is considered an important contributing factor leading to the progression of the disease.

DETAILED DESCRIPTION:
Osteoarthritis is the most common type of disease that results from an abnormality in joint function. Osteoarthritis(OA) is a condition that is characterized by progressive loss of articular cartilage of a joint and causes pain. Yamda et al. found that the strength of hip adductors increases with the severity of the disease. This reflects that more use of these muscles lower knee adductor moment 54. Considering this research, knee loads can be altered by strengthening hip muscles. Pakistan is listed in 3rd world countries and the poverty index is high. Many patients show reluctance in going to clinics for the physiotherapeutic management of knee OA. So, the present research intends to investigate the effects of home-based hip strengthening exercise on pain, functions, and range of motion in elderly knee osteoarthritis patients.

ELIGIBILITY:
Inclusion Criteria:

* The age group was from 40 to 60 years.
* Both males and females were included.
* Average knee pain on walking >3 on an 11-point scale (NPRS) (0 no pain; 10 maximal pain).
* participants can walk independently without any assistive devices
* Diagnosed patients of grade II & III of Kallgren and Lawrence scale for knee osteoarthritis referred by an orthopaedic surgeon

Exclusion Criteria:

* History of osteoporosis.
* Leg length discrepancy or structural deformity
* Knee surgery or TKR.
* Corticosteroid injection in knee joint
* Systemic arthritic condition
* History of tibiofemoral and patellofemoral replacement
* Any other neurological and muscular condition affecting the lower limb
* Any history of radiculopathy.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
intensity of Pain | baseline data
  The numerical Pain Rating Scale will be used to measure pain.
intensity of Pain | at the end of 6th week
  The numerical Pain Rating Scale will be used to measure pain.
Range of Motion | baseline data
  A goniometer will be used to measure a range of motion.
Range of Motion | at the end of 6th week
  A goniometer will be used to measure a range of motion.
Functional Disability | baseline data
  KOOS Scale will be used to measure functional disability.
Functional Disability | at the end of 6th week
  KOOS Scale will be used to measure functional disability.

CONTACTS AND LOCATIONS:
Overall Officials: faizan asghar, Principal Investigator — University of Lahore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valdes AM, McWilliams D, Arden NK, Doherty SA, Wheeler M, Muir KR, Zhang W, Cooper C, Maciewicz RA, Doherty M. Involvement of different risk factors in clinically severe large joint osteoarthritis according to the presence of hand interphalangeal nodes. Arthritis Rheum. 2010 Sep;62(9):2688-95. doi: 10.1002/art.27574. PMID 20499385
- [Background] Blagojevic M, Jinks C, Jeffery A, Jordan KP. Risk factors for onset of osteoarthritis of the knee in older adults: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2010 Jan;18(1):24-33. doi: 10.1016/j.joca.2009.08.010. Epub 2009 Sep 2. PMID 19751691
- [Background] Fatima S, Arslan SA, Sharif F, Ahmad A, Gillani SA, Zaheer A. Translation, cross-cultural adaptation and psychometric properties of the Urdu version of knee injury and osteoarthritis outcome score questionnaire for Pakistani population. BMC Musculoskelet Disord. 2021 Jun 26;22(1):592. doi: 10.1186/s12891-021-04477-1. PMID 34174864
- [Result] Bhatia D, Bejarano T, Novo M. Current interventions in the management of knee osteoarthritis. J Pharm Bioallied Sci. 2013 Jan;5(1):30-8. doi: 10.4103/0975-7406.106561. PMID 23559821
- [Result] Farrokhi S, Voycheck CA, Tashman S, Fitzgerald GK. A biomechanical perspective on physical therapy management of knee osteoarthritis. J Orthop Sports Phys Ther. 2013 Sep;43(9):600-19. doi: 10.2519/jospt.2013.4121. PMID 23756435
- [Result] Safran-Norton CE, Sullivan JK, Irrgang JJ, Kerman HM, Bennell KL, Calabrese G, Dechaves L, Deluca B, Gil AB, Kale M, Luc-Harkey B, Selzer F, Sople D, Tonsoline P, Losina E, Katz JN. A consensus-based process identifying physical therapy and exercise treatments for patients with degenerative meniscal tears and knee OA: the TeMPO physical therapy interventions and home exercise program. BMC Musculoskelet Disord. 2019 Nov 4;20(1):514. doi: 10.1186/s12891-019-2872-x. PMID 31684921
- [Result] Arhos EK, Thoma LM, Grindem H, Logerstedt D, Risberg MA, Snyder-Mackler L. Association of Quadriceps Strength Symmetry and Surgical Status With Clinical Osteoarthritis Five Years After Anterior Cruciate Ligament Rupture. Arthritis Care Res (Hoboken). 2022 Mar;74(3):386-391. doi: 10.1002/acr.24479. Epub 2022 Jan 19. PMID 33026698